CLINICAL TRIAL: NCT06114251
Title: Hepatitis B Virus Reactivation: a Cautionary Event After Liver Transplantation for Patients With Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT2023-ZJU-OBS2
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First Affiliated Hospital, Zhejiang University School of Medicine
  Interventions: Diagnostic Test: Diagnosis of postoperative recurrence of liver cancer
- Shulan (Hangzhou) Hospital
  Interventions: Diagnostic Test: Diagnosis of postoperative recurrence of liver cancer

INTERVENTIONS:
Diagnostic Test: Diagnosis of postoperative recurrence of liver cancer — HBV serological markers, such as hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg) and HBV DNA were monitored regularly. The alpha-fetoprotein (AFP) level was determined every 1-2 months. The ultrasound or computed tomography or magnetic resonance imaging was performed every 3-6 months in HCC patients who underwent liver transplantation.

SUMMARY:
Highly active hepatitis B virus (HBV) is known to be associated with poor outcomes in patients with hepatocellular carcinoma (HCC). This study aims to investigate the relationship between HBV status and HCC recurrence after liver transplantation. The study retrospectively analyzed HCC patients undergoing liver transplantation in 2 centers between January 2015 and December 2020. We reviewed post-transplant HBV status and its association with outcomes.

ELIGIBILITY:
Inclusion Criteria:

* (1) preoperative diagnosis of HBV-related HCC and (2) pathologically confirmed HCC.

Exclusion criteria

* (1) non-HBV-related HCC; (2) simultaneous presence of other tumors; (3) re-transplantation; (4) presence of portal vein tumor thrombus; and (5) a survival time of less than 90 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2015 to December 2020, the electronic medical records of liver cancer patients who underwent liver transplantation at the First Affiliated Hospital, Zhejiang University School of Medicine and Shulan (Hangzhou) Hospital were retrospectively reviewed.Recipients were followed up after liver transplantation until Dec 31, 2022. During the follow-up period, the recipients were managed according to a standard protocol. All recipients received a nucleoside analog after liver transplantation. HBV serological markers, such as hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg) and HBV DNA were monitored regularly. The alpha-fetoprotein (AFP) level was determined every 1-2 months. The ultrasound or computed tomography or magnetic resonance imaging was performed every 3-6 months in HCC patients who underwent liver transplantation.
Sampling Method: Probability Sample
Enrollment: 920 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative recurrence of liver cancer | 2015.1.1-2020.12.31

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Lu D, Chen J, Zhang J, Zhuo J, Lin Z, Cao C, Shen W, He C, Chen H, Hu Z, Sun Y, Wei X, Zhuang L, Zheng S, Xu X. Post-transplant hepatitis B virus reactivation impacts the prognosis of patients with hepatitis B-related hepatocellular carcinoma: a dual-centre retrospective cohort study in China. Int J Surg. 2024 Apr 1;110(4):2263-2274. doi: 10.1097/JS9.0000000000001141. PMID 38348848